CLINICAL TRIAL: NCT05528107
Title: Comparison of Laparoscopic Intraperitoneal Onlay Mesh (IPOM Plus) and Extended Totally Extraperitoneal (eTEP) Repair for Incisional Hernia - a Randomized Controlled Trial
Brief Title: Laparoscopic IPOM Plus vs. eTEP Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: City Clinical Hospital No.1 named after N.I. Pirogov (Other)
Collaborators: Pirogov Russian National Research Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2907-1/22
Record Dates: First submitted 2022-08-30; First posted 2022-09-06 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Incisional Hernia of Midline of Abdomen
Keywords: incisional ventral hernia; IPOM; eTEP; pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laparoscopic Intraperitoneal Onlay Mesh plus ventral hernia repair (Active Comparator): Laparoscopic Intraperitoneal Onlay Mesh plus repair will be used to perform a minimally invasive ventral hernia repair with intraperitoneal mesh placement and suturing hernia defect.
  Interventions: Procedure: Lap IPOM plus
- Extended-view totally extraperitoneal ventral hernia repair (Active Comparator): Extended-view totally extraperitoneal ventral hernia repair will be used to perform minimally invasive ventral hernia repair with retrorectus mesh placement
  Interventions: Procedure: eTEP

INTERVENTIONS:
Procedure: Lap IPOM plus — Participants will undergo Lap IPOM plus repair according to the assigned treatment arm.
  Other Names: Laparoscopic Intraperitoneal Onlay Mesh plus ventral hernia repair
  Arms: Laparoscopic Intraperitoneal Onlay Mesh plus ventral hernia repair
Procedure: eTEP — Participants will undergo eTEP repair according to the assigned treatment arm.
  Other Names: Extended-view totally extraperitoneal ventral hernia repair
  Arms: Extended-view totally extraperitoneal ventral hernia repair

SUMMARY:
The survey will compare primary and secondary outcomes of laparoscopic intraperitoneal onlay mesh (IPOM plus) and extended totally extraperitoneal (eTEP) repair for incisional hernia.

The research hypothesis is the following: patients who underwent eTEP repair may experience 30% less pain, assessed on the NRS-11 scale by the end of postoperative day 1, compared with IPOM plus procedure

DETAILED DESCRIPTION:
The use of minimally invasive surgery for the treatment of patients with incisional ventral hernias has significant advantages over open surgery. According to the current guidelines, the optimal technique for IPOM repair is a combination of suturing hernia defect and implantation an intraperitoneal anti-adhesive coated mesh prosthesis - the so-called "IPOM plus" technology (R.Bittner et al., 2019). The development of laparoscopic surgery has led to the new minimally invasive technique for ventral hernia repair - extended-view totally extraperitoneal plasty (eTEP) (I. Belyansky et al., 2018). An important advantage of eTEP is the non-fixation technique of implant placement due to correct positioning compared to the need for combined fixation for IPOM or IPOM plus, which probably affects on the level of postoperative pain in the early postoperative period.

The results of the first RCT comparing IPOM and eTEP ventral hernia repair were recently published (Mayank J. et al., 2022). It was demonstrated the benefits of eTEP repair in several aspects: less pain in the early postoperative period, as well as a faster return to physical activity and lower intervention costs. However, a significant limitation of this RCT is the analysis of interventions in a mixed group of patients with primary ventral and incisional hernias, as well as the use of IPOM procedure without suturing the hernia defect.

The sample size was determined based on the above hypothesis regarding the primary point of the study. Considering trial of Asencio F. et al. (2009) in a group of patients with incisional ventral hernias, the level of pain at the end of the first postoperative day after IPOM repair was 4.76 according to the VAS (visual analog scale) with a standard deviation of 1.975. Assuming α (type I error rate) 0.05, β 0.20, it would need a total sample size of 60 patients. Taking into account the probability of loss of patients in the evaluation of long-term results up to 20%, 72 patients will be required (36 patients per group).

Taking into account the inconsistency of the literature data on the level of pain in the early postoperative period after IPOM procedure for incisional ventral hernia repair, as well as the established primary point of the study, the investigators plan an additional calculation with correction of the sample size after evaluation intermediate results upon reaching 50% of enrolled patients of the initially established.

ELIGIBILITY:
Inclusion Criteria:

* midline incisional hernia
* defect width 2-6 cm
* ASA I-II class
* Elective hernia repair
* Considered eligible for minimally invasive ventral hernia repair
* Able to give informed consent
* Able to tolerate general anesthesia

Exclusion Criteria:

* primary ventral herna
* lateral hernia with/without midline
* defect width more than 6 cm
* refuse to give informed consent
* prior mesh placement in the retrorectus space

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2023-02-14 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
pain on postoperative day 1 | postoperative day 1
  Pain score will be assessed using the Numeric Pain Rating Scale. The mean pain score is calculated between pain values at rest and on coughing.
  Participants verbally requested to rate their pain : "Rate your pain from 0 (no pain) to 10 (unbearable pain)". 0 point is the minimum and 10 point is the maximum. The higher the score, the more severe the pain.

SECONDARY OUTCOMES:
pain on postoperative days 7 and 30 | postoperative 7 (±1) and 30 (±3) days
  Pain score will be assessed using the Numeric Pain Rating Scale. The mean pain score is calculated between pain values at rest and on physical activity.
  Participants verbally requested to rate their pain : "Rate your pain from 0 (no pain) to 10 (unbearable pain)". 0 point is the minimum and 10 point is the maximum. The higher the score, the more severe the pain.
number of participants with chronic pain | postoperative day 100 (±5 days)
  Persisted pain in surgical site more than 90 days after surgery. Pain score will be assessed using the Numeric Pain Rating Scale. Participants verbally requested to rate their pain : "Rate your pain from 0 (no pain) to 10 (unbearable pain)". 0 point is the minimum and 10 point is the maximum. The higher the score, the more severe the pain.
length of stay | 30 days after surgery
  From date of hospital admission until discharge. The length of hospital stay (days)
postoperative complications | 30 days after surgery
  Number of participants with postoperative complications, evaluated by Clavien-Dindo classification of surgical complications from Dindo et al.
analgetic consumption | 48 hours after surgery
  Consumption of analgesics during the first 48 hours after surgery
pain 6 hours after surgery | 6 hours (± 1 hour) after surgery
  Pain score will be assessed using the Numeric Pain Rating Scale. The mean pain score is calculated between pain values at rest and on coughing.
  Participants verbally requested to rate their pain : "Rate your pain from 0 (no pain) to 10 (unbearable pain)". 0 point is the minimum and 10 point is the maximum. The higher the score, the more severe the pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical City Hospital #1 named after N.I. Pirogov, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No